CLINICAL TRIAL: NCT05997576
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase 3 Study of TG103 Injection in the Management of Non-diabetic Overweight or Obesity
Brief Title: A Study of TG103 Injection in Non-diabetic Overweight or Obesity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSPC Baike (Shandong) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SYSA1803-013
Record Dates: First submitted 2023-08-08; First posted 2023-08-18 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Overweight or Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TG103 22.5 mg (Experimental): Administered subcutaneously once every week for 52 weeks. Doses gradually increased to 22.5 mg.
  Interventions: Drug: TG103 22.5 mg
- Placebo (Placebo Comparator): Administered subcutaneously once every week for 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TG103 22.5 mg — Subcutaneous injections with calorie restrict diet and increased physical activity for 52 weeks. Doses gradually increased from 7.5 mg to 22.5 mg.
  Arms: TG103 22.5 mg
Drug: Placebo — Subcutaneous injections with calorie restrict diet and increased physical activity for 52 weeks.
  Arms: Placebo

SUMMARY:
This study is a multicenter, randomized, double-blind, placebo-controlled, parallel phase 3 study to evaluate efficacy, safety, pharmacokinetics characteristics and immunogenicity of TG103 injection, a GLP-1 receptor agonist, for weight management in non-diabetic patients with BMI greater than or equal to 28 kg/m2 or greater than 24 kg/m2 in the presence of comorbidities, in addition to lifestyle intervention (calorie restrict diet and increased physical activity).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years ≤ age ≤ 75 years.
* Body Mass Index (BMI) ≥ 28 kg/m^2, or 24 kg/m^2 < BMI ≤ 28 kg/m^2 with at least one of obesity-related complications.
* Regular diet and exercise and stable body weight (i.e., self-reported body weight change < 5%) within 12 weeks before screening as well as body weight ≥ 60 kg at screening.
* Weight loss less than 5% or no weight loss after diet and exercise intervention for at least 12 weeks.
* Be able to understand the trial and complete the procedures, and be voluntary to participate in this study and sign the informed consent.

Exclusion Criteria:

* History of type 2 diabetes, type 1 diabetes or hypoglycemia.
* Overweight or obesity due to disease or drug; or weight increase due to non-fat mass increase; or monogenic obesity.
* Medications or products which are judged by investigators to cause change in weight and influence trial evaluations have been used within 12 weeks before screening or will be used during study.
* Weight loss less than 5% by monotherapy or combination with GLP-1 receptor agonists for at least 12 weeks before screening.
* Bariatric surgery within 12 months before screening; or no full recovery from any surgery or injury at screening; or gastrointestinal motility dysfunction due to gastrointestinal surgery.
* Participation in any clinical trial to receive treatment within 12 weeks before screening, or participation in clinical trial to receive TG103 before screening.
* History of allergy or suspected allergy to GLP-1 receptor agonists or antibody agents, or suspected allergy to TG103 judged by investigator due to other severe allergy history.
* Personal history or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2 (MEN-2).
* History or screening ultrasound reports of chronic pancreatitis, acute pancreatitis, etc.
* History of severe gastrointestinal disease; or gastrointestinal symptom at screening; or discontinuation of GLP-1 receptor agonist, GLP-1/GIP receptor agonist, GLP-1/GCG receptor agonist or metformin due to gastrointestinal adverse reaction.
* Severe infection at screening.
* Skin disorder that influences safety evaluation at screening.
* History of severe disease or malignant tumor.
* Systolic blood pressure ≥ 160 mmHg, diastolic blood pressure ≥ 100 mmHg, NYHA Grade Ⅲ-Ⅳ, QTc interval prolongation or severe arrhythmia at screening.
* History of abnormal thyroid function with requirement of medication treatment at screening, or screening TSH beyond the normal reference range.
* One of the followings at screening: 1) HbA1c ≥ 6.5%, or screening FPG ≥ 7.0mmol/L or<2.8mmol/L; 2) calcitonin ≥ 50 ng/L; 3) ALT or AST>3 × UNL (upper normal limit), or total bilirubin>1.5 × UNL; 4) blood amylase or lipase>1.5 × UNL, 5) TG>5.6mmol/L, 6) eGFR<60ml/min/1.73m2 , 7) positive of HBsAg, HCV-antibody, HIV-antibody or anti-TP antibody, 8) WBC< 3×10^9/L, or Hb <100g/L, 9) INR>1.2.
* History of drug abuse, drug dependence or alcoholism.
* History of moderate to severe depression, or screening Patient Health Questionaire-9 (PHQ-9) score ≥ 15.
* The fertile female who is pregnant, breast-feeding or with blood HCG positive at screening; or the fertile participants and their partner cannot use an effective contraceptive method during the trial and within 3 months after the end of treatment.
* Other situations unsuitable for this study in the investigator's opinion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 675 (Actual)
Dates: Start 2023-11-22 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with weight loss of ≥ 5% at week 40 | From baseline to week 40
  Weight loss is percentage change at week 40 compared with baseline.
Relative percentage change from baseline in body weight at week 40 | From baseline to week 40
  Weight loss is percentage change at week 40 compared with baseline.

SECONDARY OUTCOMES:
Proportion of participants with weight loss of ≥ 5% at week 52 | From baseline to week 52
  Weight loss is percentage change at week 52 compared with baseline.
Relative percentage change from baseline in body weight at week 52 | From baseline to week 52
  Weight loss is percentage change at week 52 compared with baseline.
Proportion of participants with weight loss of ≥ 10% | From baseline to week 40, 52
  Weight loss is percentage change at week 40 and week 52 compared with baseline.
Change from baseline in body weight (kg) | From baseline to week 40, 52
Change from baseline in waist circumference (cm) | From baseline to week 40, 52
Change from baseline in HbA1c (%) | From baseline to week 40, 52
Change from baseline in fasting plasma glucose (mmol/L) | From baseline to week 40, 52
Change from baseline in fasting insulin (mU/L) | From baseline to week 40, 52
Change from baseline in total cholesterol (mmol/L) | From baseline to week 40, 52
Change from baseline in triglyceride (mmol/L) | From baseline to week 40, 52
Change from baseline in low density lipoprotein cholesterol (mmol/L) | From baseline to week 40, 52
Change from baseline in high density lipoprotein cholesterol (mmol/L) | From baseline to week 40, 52
Change from baseline in systolic blood pressure (mmHg) | From baseline to week 40, 52
Change from baseline in diastolic blood pressure (mmHg) | From baseline to week 40, 52

OTHER OUTCOMES:
Number of TEAEs and SAEs assessed by CTCAE V5.0 | From baseline to week 55
Proportion of participants categorized by patient health questionnaire-9 (PHQ-9) score | From baseline to week 52
Concentration of TG103 (Ctrough) | From baseline to week 55
Proportion of anti-TG103-antibody-positive participants | From baseline to week 55
  Plasma anti-TG103 antibody will be measured at baseline to establish a positive/negative cut-off point and during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Li Yan, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Clinical Trials Information Group, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: Undecided